CLINICAL TRIAL: NCT04229576
Title: Pain Relief During Unsedated Office Hysteroscopy by Applying Transcutaneous Electrical Nerve Stimulation : Randomized Controlled Trial
Brief Title: TENS Efficacy in Pain Relief During Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ebtihal Sameih Ali Alnomany, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Using TENS to relief pain during hystroscopy (Active Comparator): device intensity (amplitude) will be individually adjusted to each participant's maximum sensory level (strongest reported tingling feeling without pain and with no muscle contractions, the TENS output intensity will be increased during the treatment every time the patient accommodated to the TENS stimulus.
  Interventions: Device: TENs
- Using placebo TENS (not active) during hystroscopy (Placebo Comparator): participants will be connected to the TENS unit in exactly the same way as participants in the active TENS group with the unit emitting the active indicator light and sound but delivering no electrical stimulation.
  Interventions: Device: TENs

INTERVENTIONS:
Device: TENs — Assessing the efficacy of TENs in pain relieve during office hysteroscopy .

SUMMARY:
Pain Relief During Unsedated Office Hysteroscopy by Applying Transcutaneous Electrical Nerve Stimulation : Randomized controlled trial

DETAILED DESCRIPTION:
Patients fulfilling inclusion criteria will be distributed in two groups, each one will be (60) patients (more than sample size number) to avoid the drop in the size of the study.

Group (A):(60) Active TENS during office hysteroscopy. Group (B)(60) placebo TENS during office hysteroscopy. The active TENS intervention consisted of a varying high-frequency (80-100 Hz), pulse duration 400-microseconds.Transcutaneous electrical nerve stimulation therapy will be initiated 5 minutes before starting the hysteroscopy and for the duration of the procedure. Two sets of two self-adhesive electrodes (circular pads) will be placed parallel to the spinal cord at the T10-L1 and S2-S4 levels .

Group (A)(60) Active TENs during office hysteroscopy The device intensity (amplitude) will be individually adjusted to each participant's maximum sensory level (strongest reported tingling feeling without pain and with no muscle contractions. Patients will be informed about the importance of maintaining the stimulation at a maximum non painful level. Thus, the TENS output intensity will be increased during the treatment every time the patient accommodated to the TENS stimulus. All the hysteroscopies will be performed by the same experienced consultant in (ECDU), who will be blinded to the patients' group allocations. Uterine cavity will be distended with normal saline

Group (B):(60) placebo TENs during office hysteroscopy To achieve blinding in the placebo group, participants will be connected to the TENS unit in exactly the same way as participants in the active TENS group with the unit emitting the active indicator light and sound but delivering no electrical stimulation.

Primary Outcome Measures :

The level of pain at the end of office hysteroscopy procedure (primary outcome) will be measured 5 minutes after procedure on a 100-mm-long horizontal line visual analog scale (VAS; 0 mm=no pain and 100 mm=worst possible pain).

A discrete, 5-point, verbal Likert scale including the following options: "no pain," "minimal pain," "moderate pain," "severe pain," and "worst pain possible," will be used to assess the internal consistency of the pain rating 5 minutes after procedure.

Secondary Outcome Measures The pain of hysteroscopy entry, contact, and biopsy. The duration of the procedure, vital parameters (blood pressure, heart rate, arterial oxygen saturation), vasovagal symptoms (dizzin ess, nausea, vomiting, shoulder pain, vertigo, sweating, or fainting), and unusual or adverse TENS events (skin allergy, pain, or burning at the electrode site) will be recorded during all the hysteroscopy procedures.

Finally, the level of satisfaction with the hysteroscopy, as indicated on a scale of ( 0-10), was measured at the end of the procedure .

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal endometrial thickening >4mm.
* Suspicious endometrial polyp or leiomyoma.
* Infertility study.
* Menstrual disorder.
* Suspicious endometrial carcinoma

Exclusion Criteria:

* • Genital infection.

  * Undiagnosed genital bleeding.
  * Contraindication to office hysteroscopy.
  * Previous cervical surgery.
  * Neurological deficit.
  * Chronic or preprocedural use of opioids or psychoactive drugs.
  * Previous experience in TENS.
  * Cutaneous damage on the application sites.
  * Pacemakers or automatic implanted cardiac defibrillators.
  * Refusal to sign the informed consent form.
  * Inability to understand informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Level of pain:visual analog scale | 5 minutes after procedures
  Using visual analog scale VAS; 0 mm=no pain and 100 mm=worst possible pain).
Verbal likert scale | 5 minutes after procedures
  A discrete, 5-point, verbal Likert scale including the following options: "no pain," "minimal pain," "moderate pain," "severe pain," and "worst pain possible," was also used to assess the internal consistency of the pain rating within the study.

SECONDARY OUTCOMES:
Pain during procedures | 5 minutes after procedures
  The pain of hysteroscopy entry, contact, and biopsy.
The duration of procedures | 5 minutes after procedures
  The duration of procesures
vital parameters | 5 minutes after procedures
  Blood pressure
Vital parameters | 5 minutes after procedures
  Heart rate
Vital parameters | 5 minutes after saturation
  Arterial oxygen saturation
Vasovagal symptoms | 5 minutes after procedures
  vasovagal symptoms (dizziness, nausea, vomiting, shoulder pain, vertigo, sweating, or fainting)
TENS advers effect | 5 minutes after procedures
  unusual or adverse TENS events (skin allergy, pain, or burning at the electrode site) will be recorded during all the hysteroscopy procedures.
Level of satisfaction | 5 minutes after procedures
  Finally, the level of satisfaction with the hysteroscopy, as indicated on a scale of ( 0-10), was measured at the end of the procedure .

CONTACTS AND LOCATIONS:
Overall Officials: Ebtihal Sa Ali, Principal Investigator — Ain Shams University
Locations (1):
- Ebtihal Sameih Ali Alnomany, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All primary and secondery outcomes will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Completed study
Access Criteria: Data access will be reviewed by an external independant review panel. Requests will be required to sign a data access agreement